CLINICAL TRIAL: NCT05370599
Title: Hypertension in Young Adults Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding limitations.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 21-35626
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: 3x3 by BP agent and BP monitoring approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (9):
- Amlodipine 2.5 mg + Home BP monitoring with cuffed device (Active Comparator): Use of at least the minimum dose of amlodipine and use of a home BP monitoring device for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: amlodipine; Device: Home BP monitoring with cuffed device
- Chlorthalidone 12.5 mg + Home BP monitoring with cuffed device (Experimental): Use of at least the minimum dose of chlorthalidone and use of a home BP monitoring device for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: Chlorthalidone; Device: Home BP monitoring with cuffed device
- Losartan 12.5 mg daily + home BP monitoring with cuffed device (Experimental): Use of at least the minimum dose of losartan and use of a home BP monitoring cuffed device only for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: Losartan; Device: Home BP monitoring with cuffed device
- amlodipine 2.5 mg daily + home BP monitoring with patch (Experimental): Use of at least the minimum dose of this agent and use of a home BP monitoring device only + a patch for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: amlodipine; Device: Home BP monitoring with cuffed device + BP patch
- Chlorthalidone 12.5 mg daily + home BP monitoring with patch (Experimental): Use of at least the minimum dose of this agent and use of a home BP monitoring device only + a patch for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: Chlorthalidone; Device: Home BP monitoring with cuffed device + BP patch
- Losartan 12.5 mg daily + home BP monitoring with patch (Experimental): Use of at least the minimum dose of this agent and use of a home BP monitoring device only + a patch for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: Losartan; Device: Home BP monitoring with cuffed device + BP patch
- amlodipine 2.5 mg daily + home BP monitoring with watch (Experimental): Use of at least the minimum dose of this agent and use of a home BP monitoring device only + a watch for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: amlodipine; Device: Home BP monitoring with cuffed device + BP watch
- chlorthalidone 12.5 mg daily + home BP monitoring with watch (Experimental): Use of at least the minimum dose of this agent and use of a home BP monitoring device only + a watch for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: Chlorthalidone; Device: Home BP monitoring with cuffed device + BP watch
- losartan 12.5 mg daily + home BP monitoring with watch (Experimental): Use of at least the minimum dose of this agent and use of a home BP monitoring device only + a watch for BP monitoring
  Interventions: Drug: Anti-hypertensive agent: Losartan; Device: Home BP monitoring with cuffed device + BP watch

INTERVENTIONS:
Drug: Anti-hypertensive agent: amlodipine — Patients with hypertension will be randomly assigned to be treated with amlodipine, chlorthalidone, or losartan. All drugs will be initiated at the lowest dose and uptitrated as needed to achieve standard BP targets.
  Arms: Amlodipine 2.5 mg + Home BP monitoring with cuffed device; amlodipine 2.5 mg daily + home BP monitoring with patch; amlodipine 2.5 mg daily + home BP monitoring with watch
Drug: Anti-hypertensive agent: Chlorthalidone — Patients with hypertension will be randomly assigned to be treated with amlodipine, chlorthalidone, or losartan. All drugs will be initiated at the lowest dose and uptitrated as needed to achieve standard BP targets.
  Arms: Chlorthalidone 12.5 mg + Home BP monitoring with cuffed device; Chlorthalidone 12.5 mg daily + home BP monitoring with patch; chlorthalidone 12.5 mg daily + home BP monitoring with watch
Drug: Anti-hypertensive agent: Losartan — Patients with hypertension will be randomly assigned to be treated with amlodipine, chlorthalidone, or losartan. All drugs will be initiated at the lowest dose and uptitrated as needed to achieve standard BP targets.
  Arms: Losartan 12.5 mg daily + home BP monitoring with cuffed device; Losartan 12.5 mg daily + home BP monitoring with patch; losartan 12.5 mg daily + home BP monitoring with watch
Device: Home BP monitoring with cuffed device — Patients will be randomized to monitor their blood pressure either with a BP cuffed device alone, versus with either or use of a BP monitoring patch or BP monitoring watch.
  Arms: Amlodipine 2.5 mg + Home BP monitoring with cuffed device; Chlorthalidone 12.5 mg + Home BP monitoring with cuffed device; Losartan 12.5 mg daily + home BP monitoring with cuffed device
Device: Home BP monitoring with cuffed device + BP patch — Patients will be randomized to monitor their blood pressure either with a BP cuffed device alone, versus with either or use of a BP monitoring patch or BP monitoring watch.
  Arms: Chlorthalidone 12.5 mg daily + home BP monitoring with patch; Losartan 12.5 mg daily + home BP monitoring with patch; amlodipine 2.5 mg daily + home BP monitoring with patch
Device: Home BP monitoring with cuffed device + BP watch — Patients will be randomized to monitor their blood pressure either with a BP cuffed device alone, versus with either or use of a BP monitoring patch or BP monitoring watch.
  Arms: amlodipine 2.5 mg daily + home BP monitoring with watch; chlorthalidone 12.5 mg daily + home BP monitoring with watch; losartan 12.5 mg daily + home BP monitoring with watch

SUMMARY:
This is a pilot randomized controlled trial which will test the effect of 3 different anti-hypertensive agents and 3 different strategies of engaging young adults in home blood pressure monitoring on blood pressure control, with secondary outcomes focused on quality of life and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Diagnosis of hypertension or receiving anti-hypertensive therapy OR Has clinical BP readings >130/80 mmHg that would meet the definition of hypertension and have home BP readings >=125/80 mmHg

Exclusion Criteria:

* are or are planning to become pregnant, due to inability to take multiple classes of anti- hypertensive agents
* are marginally housed, due to concerns regarding routine follow-up
* are actively participating in a different interventional trial that may affect blood pressure
* are unwilling to consent to participate
* institutionalized individuals or prisoners
* are actively abusing illicit drugs or alcohol
* have a history of poor or doubtful compliance (e.g., frequently missed appointments)
* have cognitive impairment prohibiting participation in the study
* History of allergy to any of the randomized medications
* Serum potassium >5.5 meq/L at the screening visit
* BP > 160/100 mmHg in clinic (stage II hypertension), regardless of whether patient is on therapy
* eGFR < 30 mL/min/1.73 m2

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Achieved systolic blood pressure | Month 6
  Systolic blood pressure will be collected using at home cuffed devices. The readings at end of the pilot trial (or most recent readings available) will be used for analysis of the primary outcome.

SECONDARY OUTCOMES:
Adherence to home BP monitoring | Between month 0 and 6
  Percent of weeks with at least 9 self-measured readings per week

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Ku, MD MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson HM, Warner RC, Bartels CM, LaMantia JN. "They're younger... it's harder." Primary providers' perspectives on hypertension management in young adults: a multicenter qualitative study. BMC Res Notes. 2017 Jan 3;10(1):9. doi: 10.1186/s13104-016-2332-8. PMID 28057065